CLINICAL TRIAL: NCT02681913
Title: The Effect of Adenosine on Myocardial Protection in Intermittent Warm Blood Cardioplegia: A Randomized Placebo-controlled Trial
Brief Title: Adenosine as an Adjunct to Blood Cardioplegia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amphia Hospital (Other)
Responsible Party: Principal Investigator, Jeffrey Engelhart, PharmD, MSc, Amphia Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1437; 2015-001923-22 (EudraCT Number)
Record Dates: First submitted 2016-02-03; First posted 2016-02-15 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Pathological Processes; Cardiomyopathies
Keywords: Cardioplegia; Cardiac Surgery; Adenosine; Therapeutic Uses; Intermittent warm blood cardioplegia; Minimally Invasive Surgery; minimally invasive mitral valve plasty (mini-MPL); minimally invasive mitral valve replacement (mini-MVR)
MeSH Terms: conditions — Pathologic Processes; Cardiomyopathies | interventions — Adenosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard cardioplegia (No Intervention): Delivery of cardioplegic solutions will be according to the standard protocol (Amphia hospital, Breda, the Netherlands). Oxygenated blood and cardioplegic maintenance solution is delivered in a 20:1 ratio. Cardioplegic solutions will be administered at 20-minutes intervals. The flow of the cardioplegia must be at 300 ml/min, the duration is approximately 1 minute.
  The cardioplegic maintenance solution consists of a 500 ml normal saline (0.9% NaCl) infusion bag. Potassiumchloride (20 mmol) and magnesiumsulphate (1000 mg) is added according to standard protocol.
  This arms receives standard intermittent 20:1 diluted warm blood cardioplegic solution.
  Intervention: n/a
- adenosine enriched cardioplegia (Experimental): Delivery of cardioplegic solutions will be according to the standard protocol (Amphia hospital, Breda, the Netherlands). Oxygenated blood and cardioplegic maintenance solution is delivered in a 20:1 ratio. Cardioplegic solutions will be administered at 20-minutes intervals. The flow of the cardioplegia must be at 300 ml/min, the duration is approximately 1 minute.
  The cardioplegic maintenance solution consists of a 1000 mg = 500 ml adenosine infusion bag (2 mg/ml). Potassiumchloride (20 mmol) and magnesiumsulphate (1000 mg) is added according to standard protocol.
  This arms receives adenosine enriched, intermittent 20:1 diluted warm blood cardioplegic solution.
  Intervention: Drug: Adenosine
  Interventions: Drug: Adenosine

INTERVENTIONS:
Drug: Adenosine — This group receives intermittent warm blood cardioplegia enriched with adenosine
  Other Names: Adenocor
  Arms: adenosine enriched cardioplegia

SUMMARY:
Myocardial protection is a major issue in cardiac surgery, since inadequate protection increases the risk of postoperative cardiac dysfunction. The main principle of myocardial protection in cardiac surgery is to preserve myocardial function by preventing ischemia with blood cardioplegia . Previous studies have shown that adenosine as an adjunct to blood cardioplegia can be safely used in cardiac surgery. In the Amphia Hospital, adenosine is already used as standard care as an initial cardioplegic bolus in minimally invasive port access operations. Whether, adenosine as an adjunct to intermittent warm blood cardioplegia, has an added value remains unclear. Therefore the investigators would like to investigate the effect of the addition of adenosine to standard intermittent warm blood cardioplegia in patients scheduled for minimally invasive, port access operations (mitral valve surgery).

Half of the participants will receive standard intermittent warm blood cardioplegia, while the other half will receive intermittent warm blood cardioplegia enriched with adenosine.

DETAILED DESCRIPTION:
Myocardial protection is a major issue in cardiac surgery, since inadequate protection increases the risk of postoperative cardiac dysfunction. The main principle of myocardial protection in cardiac surgery is to preserve myocardial function by preventing ischemia with blood cardioplegia . Previous studies have shown that adenosine as an adjunct to blood cardioplegia can be safely used in cardiac surgery. In the Amphia Hospital, adenosine is already used as standard care as an initial cardioplegic bolus in minimally invasive port access operations. Whether, adenosine as an adjunct to intermittent warm blood cardioplegia, has an added value remains unclear. Therefore the investigators would like to investigate whether the addition of adenosine to standard intermittent warm blood cardioplegia reduces the 6-hours post-operative cardiac troponin T (cTnT) in patients scheduled for minimally invasive, port access operations (mitral valve surgery).

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgical patients

  * minimally invasive, port access surgery (mitral valve surgery)

Exclusion Criteria:

* All non-minimally invasive, port access surgery
* Theophylline or dipyridamole use up to 24 hours prior to surgery
* Products that contain caffeine of theobromine up to 12 hours prior to surgery (coffee, chocolate, energizing drinks (e.g. Red Bull), tea, soda (coke), etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
6-hour cardiac Troponin T (cTnT) release | 6 hours post-operative
  The primary end point is 6-hour cTnT release

SECONDARY OUTCOMES:
18-hour cardiac Troponin T (cTnT) area under the curve (AUC) release | cardiac Troponin T (cTnT) AUC will be assessed at different time points, the latest up to 18 hours after ICU arrival
  18-hour postoperative AUC release of cardiac troponin T Routine blood samples pre-operatively from peripheral blood (T0); post-operatively, from peripheral blood, at arrival at ICU (T1) and 6 hours after arrival at ICU (T2), and 18 hours after arrival at ICU (T3).
Incidence of myocardial injury on 12-lead ECG | participants will be followed for the duration of ICU stay, an expected average of 2 days
  Incidence of myocardial injury on 12-lead ECG
  * New-onset Left bundle branch block (LBBB)
  * New-onset Q wave
Vasoactive-inotropic score | participants will be followed for the duration of ICU stay, an expected average of 2 days
  The hourly doses of the following inotropic and vasoactive medications are recorded for the first 18 h after post-operative admission to the ICU: dopamine, dobutamine, epinephrine, norepinephrine, milrinone and vasopressin.
Vasoconstrictor usage | participants will be followed for the duration of ICU stay, an expected average of 2 days
  Vasoconstrictor usage yes/no
Incidence of new onset Atrial fibrillation (AF) | participants will be followed for the duration of ICU stay, an expected average of 2 days
  Incidence of new onset AF
Routine blood samples | Routine blood samples will be assessed at different time points, the latest up to 6 hours after ICU arrival
  The amount of creatine kinase MB (CK-MB) and Creatinine at different time intervals. preoperatively from peripheral blood (T0); post-operatively, from peripheral blood, at arrival at ICU (T1) and 6 hours after arrival at ICU (T2)
Mean arterial pressure (MAP) | participants will be followed for the duration of ICU stay, an expected average of 2 days
  Haemodynamic monitoring
postoperative left ventricular ejection fraction (LVEF) | postoperative after skin closure, an expected average of 3 hours after starting surgery
  3-D transesophageal echocardiography (TEE) postoperative left ventricular ejection fraction (LVEF) after skin closure
Wall Motion Score Index (WMSI) | postoperative after skin closure, an expected average of 3 hours after starting surgery
  3-D transesophageal echocardiography (TEE) Wall Motion Score Index (WMSI) after skin closure
Heart rate (HR) | participants will be followed for the duration of ICU stay, an expected average of 2 days
  Haemodynamic monitoring. Heart rate will be measured in beats per minute (bpm).
Cardiac index (CI) | participants will be followed for the duration of ICU stay, an expected average of 2 days
  Cardiac index (CI) is a haemodynamic parameter that relates the cardiac output (CO) from left ventricle in one minute to body surface area (BSA)
Systemic vascular resistance index (SVRI) | participants will be followed for the duration of ICU stay, an expected average of 2 days
  SVRI = 80 x (MAP - RAP)/CI MAP = Mean Arterial Pressure (mmHg) RAP = Right Arterial Pressure (mmHg) CI = Cardiac Index (L/min/m2)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Engelhart, PharmD, Principal Investigator — Amphia Hospital
Locations (1):
- Amphia Hospital, Breda, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahlsson A, Sobrosa C, Kaijser L, Jansson E, Bomfim V. Adenosine in cold blood cardioplegia--a placebo-controlled study. Interact Cardiovasc Thorac Surg. 2012 Jan;14(1):48-55. doi: 10.1093/icvts/ivr027. Epub 2011 Nov 15. PMID 22108937
- [Background] Cohen G, Feder-Elituv R, Iazetta J, Bunting P, Mallidi H, Bozinovski J, Deemar C, Christakis GT, Cohen EA, Wong BI, McLean RD, Myers M, Morgan CD, Mazer CD, Smith TS, Goldman BS, Naylor CD, Fremes SE. Phase 2 studies of adenosine cardioplegia. Circulation. 1998 Nov 10;98(19 Suppl):II225-33. PMID 9852907
- [Background] Cohen G, Borger MA, Weisel RD, Rao V. Intraoperative myocardial protection: current trends and future perspectives. Ann Thorac Surg. 1999 Nov;68(5):1995-2001. doi: 10.1016/s0003-4975(99)01026-7. PMID 10585118
- [Background] Chauhan S, Wasir HS, Bhan A, Rao BH, Saxena N, Venugopal P. Adenosine for cardioplegic induction: a comparison with St Thomas solution. J Cardiothorac Vasc Anesth. 2000 Feb;14(1):21-4. doi: 10.1016/s1053-0770(00)90050-8. PMID 10698387
- [Background] Mentzer RM Jr, Birjiniuk V, Khuri S, Lowe JE, Rahko PS, Weisel RD, Wellons HA, Barker ML, Lasley RD. Adenosine myocardial protection: preliminary results of a phase II clinical trial. Ann Surg. 1999 May;229(5):643-9; discussion 649-50. doi: 10.1097/00000658-199905000-00006. PMID 10235522
- [Background] Onorati F, Santini F, Dandale R, Ucci G, Pechlivanidis K, Menon T, Chiominto B, Mazzucco A, Faggian G. "Polarizing" microplegia improves cardiac cycle efficiency after CABG for unstable angina. Int J Cardiol. 2013 Sep 10;167(6):2739-46. doi: 10.1016/j.ijcard.2012.06.099. Epub 2012 Jul 12. PMID 22795715
- [Background] Jakobsen O, Naesheim T, Aas KN, Sorlie D, Steensrud T. Adenosine instead of supranormal potassium in cardioplegia: it is safe, efficient, and reduces the incidence of postoperative atrial fibrillation. A randomized clinical trial. J Thorac Cardiovasc Surg. 2013 Mar;145(3):812-8. doi: 10.1016/j.jtcvs.2012.07.058. Epub 2012 Sep 7. PMID 22964356
- [Background] Liu R, Xing J, Miao N, Li W, Liu W, Lai YQ, Luo Y, Ji B. The myocardial protective effect of adenosine as an adjunct to intermittent blood cardioplegia during open heart surgery. Eur J Cardiothorac Surg. 2009 Dec;36(6):1018-23. doi: 10.1016/j.ejcts.2009.06.033. Epub 2009 Aug 15. PMID 19683936